CLINICAL TRIAL: NCT00435643
Title: Improvement in Hypothalamic-Pituitary-Adrenal Axis Function After Continuous Positive Airway Pressure Therapy in Obstructive Sleep Apnea Syndrome
Brief Title: Influence of nCPAP on Metabolic Consequences Associated With OSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12383
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Obstructive Sleep Apnea Syndrome; Obesity
Keywords: Sleep apnea,; adiponectin ,; HPA axis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Active Comparator): 10 patients with severe OSAS (Apnea Hypopnea Index of more than 30 events per hour of sleep) were treated with nCPAP for three months and all mentioned measurements above were repeated.
  Interventions: Procedure: nasal continuous positive airway pressure

INTERVENTIONS:
Procedure: nasal continuous positive airway pressure — After an average interval of three months, 10 patients with severe OSAS (AHI of more than 30 events per hour of sleep) treated with a mean nCPAP pressure of 11.2 ± 0.7 cm of H2O were reassessed and all mentioned measurements above were repeated

SUMMARY:
Context: Obstructive sleep apnea syndrome (OSAS) is associated with cardiovascular morbidity. Recurrent episodes of occlusion of upper airways during sleep result in hormonal changes that may predispose to high cardiovascular risk.These risks can rapidly be reduced by effective nasal continuous positive airway pressure (nCPAP) therapy Objective: To evaluate hypothalamic pituitary adrenal axis, insulin resistance, blood pressure values and adipokines in severe obese patients with and without OSAS and to determine if continuous positive airway pressure therapy (nCPAP) influenced responses.

DETAILED DESCRIPTION:
Background: There is evidence that obstructive sleep apnea syndrome (OSAS) increases the risk of cardiovascular events. Sympathetic nervous system and hypothalamic-pituitary-adrenal (HPA) axis activation may be the mechanism of this relationship. We evaluate HPA axis and metabolic consequences in obese patients with and without OSAS and we determine if continuous positive airway pressure therapy (nCPAP) influenced responses.

Methods: Plasma inflammatory cytokines, insulin resistance index, 24-hour ambulatory blood pressure monitoring and overnight cortisol suppression test with 0.25 mg of dexamethasone were performed in 22 severe obese patients with OSAS and 23 obese controls. Ten patients with severe apnea were re-evaluated three months after nCPAP therapy.

Results: Body mass index, abdominal circumference, blood pressure levels and insulin resistance indexes of OSAS patients and obese controls were very similar. In OSAS patients, adiponectin (p<0.05) and salivary cortisol suppression pos DEX (p<0.05) were lower, while heart rate (p<0.05) and TNF-alpha levels (p<0.05) were higher compared with obese controls. After nCPAP therapy, patients showed a reduction in heart rate (p=0.036) and a higher cortisol suppression after dexamethasone (p=0.001) and there were no differences in insulin resistance (HOMA p=0.139), arterial blood pressure (p=0.183) and adipokines compared with baseline. Cortisol suppression was positively correlated with the improvement of apnea hypopnea index while on nCPAP therapy (r= 0.799, p=0.010).

Conclusions: Patients with OSAS present nocturnal hypercortisolism, hyperactivity of sympathetic central nervous system, a higher degree of inflammation and hypoadiponectinemia independent of the body mass index. Furthermore, hyperactivity of HPA axis and sympathetic nervous system are recovered by nCPAP.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 years
* Body mass index between 35-60 who were submitted to polysomnography

Exclusion Criteria:

* History of smoking
* Sleep apnea treatment
* Cardiovascular disease
* Malignancies tumor
* Thyroid disorders
* Depression
* Subjects with known diabetes mellitus on medications
* Chronic renal or hepatic failure
* On hormonal replacement therapy, as well as use of medication that could potentially affect steroid hormone or cytokines secretion (alcohol, psychotropics, steroids, sympathomimetics, beta-blockers).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-10; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To explore the interactive mechanisms of HPA axis, sympathetic nervous system activation, inflammatory cytokines, insulin resistance and hypertension in patients with and without sleep apnea, excluding the interference of the degree of fat accumulation. | one day

SECONDARY OUTCOMES:
To evaluate low-dose dexamethasone-induced cortisol suppression and circadian rhythm of cortisol secretion in severe obese patients with sleep apnea in response to treatment with continuous positive airway pressure. | three months

CONTACTS AND LOCATIONS:
Overall Officials: Gláucia Carneiro, MD, Principal Investigator — UNIFESP-EPM
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Buckley TM, Schatzberg AF. On the interactions of the hypothalamic-pituitary-adrenal (HPA) axis and sleep: normal HPA axis activity and circadian rhythm, exemplary sleep disorders. J Clin Endocrinol Metab. 2005 May;90(5):3106-14. doi: 10.1210/jc.2004-1056. Epub 2005 Feb 22. PMID 15728214
- [Background] Lanfranco F, Gianotti L, Pivetti S, Navone F, Rossetto R, Tassone F, Gai V, Ghigo E, Maccario M. Obese patients with obstructive sleep apnoea syndrome show a peculiar alteration of the corticotroph but not of the thyrotroph and lactotroph function. Clin Endocrinol (Oxf). 2004 Jan;60(1):41-8. doi: 10.1111/j.1365-2265.2004.01938.x. PMID 14678286
- [Background] Masserini B, Morpurgo PS, Donadio F, Baldessari C, Bossi R, Beck-Peccoz P, Orsi E. Reduced levels of adiponectin in sleep apnea syndrome. J Endocrinol Invest. 2006 Sep;29(8):700-5. doi: 10.1007/BF03344179. PMID 17033258
- [Background] Wolk R, Svatikova A, Nelson CA, Gami AS, Govender K, Winnicki M, Somers VK. Plasma levels of adiponectin, a novel adipocyte-derived hormone, in sleep apnea. Obes Res. 2005 Jan;13(1):186-90. doi: 10.1038/oby.2005.24. PMID 15761179
- [Background] Degawa-Yamauchi M, Moss KA, Bovenkerk JE, Shankar SS, Morrison CL, Lelliott CJ, Vidal-Puig A, Jones R, Considine RV. Regulation of adiponectin expression in human adipocytes: effects of adiposity, glucocorticoids, and tumor necrosis factor alpha. Obes Res. 2005 Apr;13(4):662-9. doi: 10.1038/oby.2005.74. PMID 15897474
- [Derived] Carneiro G, Florio RT, Zanella MT, Pradella-Hallinan M, Ribeiro-Filho FF, Tufik S, Togeiro SM. Is mandatory screening for obstructive sleep apnea with polysomnography in all severely obese patients indicated? Sleep Breath. 2012 Mar;16(1):163-8. doi: 10.1007/s11325-010-0468-7. Epub 2011 May 29. PMID 21626286